CLINICAL TRIAL: NCT06943339
Title: Effects of Different Compositions of Enteral Nutrition Products on Malnutrition and Biochemical Parameters
Brief Title: Impact of Enteral Nutrition Variants on Malnutrition and Biochemical Markers
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Collaborators: Sanliurfa Mehmet Akif Inan Education and Research Hospital (Other)
Responsible Party: Principal Investigator, HAKAN TOĞUÇ, Assistant professor, Inonu University
Other Study IDs: Inonu-NAD-HT-01
Record Dates: First submitted 2025-02-27; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Malnutrition
Keywords: malnutrition; intensive care; enteral nutrition; biochemical markers
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard enteral nutrition group: Participants included in the group were those who consumed a standard enteral product (1kcal/1ml) for 15 days
  Interventions: Other: Standard enteral nutrition
- High energy and protein enteral nutrition group: Participants included in the group were those who consumed high energy and protein enteral products (1.5 kcal/1ml + protein content increased) for 15 days.
  Interventions: Other: High energy and protein enteral nutrition

INTERVENTIONS:
Other: Standard enteral nutrition — It will include the baseline and 15-day follow-up data of the patients in the standard enteral nutrition group for standard product (1kkal/1ml) intake. No intervention will be made by the researchers during the treatment process of the patients.
  Groups: Standard enteral nutrition group
Other: High energy and protein enteral nutrition — It will include the baseline and 15-day follow-up data of the patients in the high energy and protein enteral nutrition group for the intake of high energy and protein containing product (1.5kkal/1ml + protein content increased). No intervention will be made by the researchers during the treatment process of the patients.
  Groups: High energy and protein enteral nutrition group

SUMMARY:
This study aims to investigate the effects of consumption of enteral nutrition products with different compositions on malnutrition and biochemical parameters in intensive care unit patients.

DETAILED DESCRIPTION:
Malnutrition is a common health problem, especially in individuals with chronic diseases, significantly decreases the quality of life and increases morbidity and mortality rates. Nutritional support plays a vital role in the prevention and treatment of malnutrition. Enteral nutrition, which is preferred especially in cases where oral nutrition is inadequate, is a frequently used method to ensure that patients receive sufficient amounts of energy and essential nutrients. The formulations of enteral nutrition products may vary according to the specific needs of the patient and the components of these products have a critical role in correcting malnutrition and improving biochemical parameters. However, studies on the efficacy of enteral products with different ingredients and their relationship with biochemical parameters in individuals at risk of malnutrition are very limited. This study aims to investigate the effects of enteral nutrition products with various compositions on malnutrition and biochemical parameters in intensive care unit patients.

This study is an observational and quasi-experimental study conducted in the Intensive Care Unit of Mehmet Akif Inan Training and Research Hospital. Inclusion criteria included being 18 years of age or older, receiving enteral nutrition during the study period (15 days) and having complete patient records. Exclusion criteria were receiving parenteral nutrition before starting enteral nutrition, patients with gastrointestinal problems contraindicating enteral nutrition, and patients who died within 15 days after starting enteral nutrition or whose formula changed. Within the scope of the research, it was planned to reach a total of 50 participants, 25 in each group. At the end of the research, 43 participants who received standard products (1kkal/1ml) and 30 participants who received products containing high energy and protein (1.5 kkal/1ml + protein content increased) were reached.

Patients included in the study design will be divided into two groups. One group will include the data of the participants receiving the standard product (1kkal/1ml) and the other group will include the data of the participants receiving the product containing high energy and protein (1.5 kkal/1ml + protein content increased). No intervention will be made by the researchers during the treatment process of the patients, only the nutritional status of the patients at the beginning of enteral nutrition and 15 days later (NRS-2002 (Nutritional Risk Score-2002), Prognostic nutrition index (PNI) and modified Glasgow prognostic score (mGPS)) and biochemical parameters will be evaluated.

NRS-2002: This scale is designed to assess risk factors associated with the patient's nutritional status and disease severity. The NRS-2002 is administered on admission and has the feature of adding an additional risk score for individuals over 70 years of age. The scale calculates a nutritional risk score based on objective criteria including the patient's body mass index, changes in dietary intake and severity of disease. The presence of malnutrition is defined when the scale score is 3 and above.

Prognostic nutrition index (PNI): This index, calculated with serum albumin level and total lymphocyte count factors, is scored by combining nutritional and immunological parameters. While albumin is an indicator of protein adequacy and nutritional status in the body, lymphocyte count reflects the immunological status of the body. A total score below 45 points is considered at risk for malnutrition and immunosuppression.

modified Glasgow prognostic score (mGPS)): This index, calculated on the basis of C-reactive protein (CRP) and albumin levels, represents a survival prognosis.

Biochemical results: Biochemical parameters such as glucose, albumin, CRP, haemoglobin, urea, creatinine, lymphocytes, leukocytes, monocytes, neutrophils, eosinophils, basophils will be recorded from patient files.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Receiving enteral nutrition during the study period (15 days)
* Having complete patient records

Exclusion Criteria:

* Receiving parenteral nutrition before starting enteral nutrition
* Patients with gastrointestinal problems contraindicating enteral nutrition
* Patients who died within 15 days after starting enteral nutrition or whose formula changed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age receiving enteral nutrition who were treated in the Intensive Care Unit of Mehmet Akif Inan Training and Research Hospital were included.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum Glucose Level (mg/dL) | Baseline and after 15 days
  Change in fasting blood glucose levels (mg/dL) from baseline to Day 15.
Change in Serum Albumin Level (g/dL) | Baseline and after 15 days
  Change in serum albumin concentration (g/dL) from baseline to Day 15.
Change in Serum CRP Level (mg/L) | Baseline and after 15 days
  Change in C-reactive protein levels (mg/L) from baseline to Day 15.
Change in Hemoglobin Level (g/dL) | Baseline and after 15 days
  Change in hemoglobin concentration (g/dL) from baseline to Day 15.
Change in Serum Urea Level (mg/dL) | Baseline and after 15 days
  Change in serum urea levels (mg/dL) from baseline to Day 15.
Change in Serum Creatinine Level (mg/dL) | Baseline and after 15 days
  Change in serum creatinine levels (mg/dL) from baseline to Day 15.
Change in Lymphocyte Count (10^3/µL) | Baseline and after 15 days
  Change in absolute lymphocyte count (10^3/µL) from baseline to Day 15.
Change in Leukocyte Count (10^3/µL) | Baseline and after 15 days
  Change in total leukocyte count (10^3/µL) from baseline to Day 15.
Change in Monocyte Count (10^3/µL) | Baseline and after 15 days
  Change in absolute monocyte count (10^3/µL) from baseline to Day 15.
Change in Neutrophil Count (10^3/µL) | Baseline and after 15 days
  Change in absolute neutrophil count (10^3/µL) from baseline to Day 15.
Change in Eosinophil Count (10^3/µL) | Baseline and after 15 days
  Change in absolute eosinophil count (10^3/µL) from baseline to Day 15.
Change in Basophil Count (10^3/µL) | Baseline and after 15 days
  Change in absolute basophil count (10^3/µL) from baseline to Day 15.

SECONDARY OUTCOMES:
Change in NRS-2002 Nutritional Risk Score | Baseline and after 15 days
  Change in NRS-2002 score, which evaluates the nutritional risk based on BMI, weight loss, food intake, and disease severity. Scores ≥3 indicate nutritional risk.
  Time Frame: Baseline and after 15 days Unit of Measure: Units on a scale (0-7)
Change in Prognostic Nutrition Index (PNI) | Baseline and after 15 days
  Change in PNI score calculated as:
  PNI=(10×SerumAlbumin[g/dL])+(0.005×TotalLymphocyteCount[/mm3])PNI = (10 × Serum Albumin [g/dL]) + (0.005 × Total Lymphocyte Count [/mm³])PNI=(10×SerumAlbumin[g/dL])+(0.005×TotalLymphocyteCount[/mm3]) Scores <45 indicate malnutrition and immunosuppression risk.
Change in Modified Glasgow Prognostic Score (mGPS) | Baseline and after 15 days
  Change in mGPS, based on CRP and albumin levels.
  Score 0: CRP ≤10 mg/L
  Score 1: CRP >10 mg/L and Albumin ≥3.5 g/dL
  Score 2: CRP >10 mg/L and Albumin <3.5 g/dL Time Frame: Baseline and after 15 days Unit of Measure: Categorical (0, 1, or 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Inan Training and Research Hospital, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data from participants were gathered solely for research objectives, adhering strictly to the ethical principles of confidentiality and protection. As such, it is not available for sharing.